CLINICAL TRIAL: NCT03724357
Title: Blood Donor CVD 9000: Collection of Blood for In Vitro Studies From Healthy Adults Who Have Received Oral Cholera Vaccine (CVD 103-HgR)
Brief Title: Blood Donor CVD 9000
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: lack of funding
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Marcelo Sztein, Assistant Professor, University of Maryland, Baltimore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HP-00082377
Record Dates: First submitted 2018-10-26; First posted 2018-10-30 (Actual); Results first posted 2023-02-02 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-01

CONDITIONS: Cholera Vaccination
MeSH Terms: interventions — Vaxchora; cholera vaccine CVD 103-HgR

STUDY DESIGN:
Intervention Model Description: Volunteers who choose to take part in this study will receive the licensed FDA-approved Oral Cholera Vaccine (Vaxchora).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Vaccination with Oral Cholera Vaccine (Vaxchora) (Experimental): Volunteers receive immunization with Vaxchora cholera vaccine. Blood draws are performed at subsequent visits.
  Interventions: Drug: Vaxchora

INTERVENTIONS:
Drug: Vaxchora — One dose. Approximately 100 mL of cold or room temperature purified bottled water is placed into a clean disposable cup. The contents of the buffer sachet are added to the water and stirred. Then the contents of the active (lyophilized vaccine) sachet are added to the water and stirred for approximately 30 seconds. The reconstituted mixture should be completely ingested within 15 minutes.
  Other Names: CVD 103-HgR

SUMMARY:
This is an open-label, non-randomized study. Volunteers will be vaccinated with the oral cholera vaccine, Vaxchora. Vaxchora has been licensed by the Food and Drug Administration (FDA) for travelers to developing countries. Volunteers will also be asked to provide blood specimens over a follow-up time period of up to eight years. The specimens obtained in this clinical research study will be used to further the investigator's understanding of the protective immunological mechanisms that can be elicited systemically and may be applicable to other enteric pathogens.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age 18 years to 64 years at the time of enrollment
* 2. Good general health as determined by a screening evaluation within 28 days before blood donation or vaccination
* 3. Provides written informed consent prior to initiation of any study procedures

Exclusion Criteria:

* 1. History of any of the following medical conditions:

  * Diabetes
  * Cancer in past 5 years (except for basal cell carcinoma of the skin and cervical carcinoma in situ)
  * Heart disease (e.g., hospitalization for a heart attack, coronary artery bypass graft, arrhythmia, or syncope, within past 5 years. Current symptoms of heart disease, such as dyspnea, angina, or orthopnea)
  * Recurrent infections (e.g., more than 3 hospitalizations for invasive bacterial infections such as pneumonia or meningitis)
  * Current drug or alcohol abuse
  * Active ulcer disease or ongoing intestinal condition
  * Treatment for anemia in last 6 months
  * Treatment with anti-malarial drugs within ten days prior to study vaccination
  * Treatment with antibiotics within 14 days prior to study vaccination
  * Immunodeficiency or immunosuppression from illness or treatment
* 2. Close contact within 7 days following study vaccination with a person who has an immunodeficiency or immunosuppression from illness or treatment
* 3. History of cholera infection or cholera vaccination
* 4. Any of the following complete blood count (CBC) abnormalities during screening:

  * white blood cells (WBC) <0.81 x lower limit of normal (LLN) or > 1.09 x upper limit of normal (ULN)
  * Hemoglobin <0.91 x LLN or >1.18 x ULN (women) or <0.92 x LLN or >1.18 x ULN (men)
  * Platelet count <0.8 x LLN or > 1.2 x ULN
* 5. Any of the following laboratory abnormalities during screening:

  * serum glutamic oxaloacetic transaminase (SGOT) or serum glutamic pyruvic transaminase (SGPT) >1.5 times normal
  * Positive serology for HIV antibody
* 6. Poor peripheral venous access for blood donation
* 7. Other condition that the opinion of the investigator would jeopardize the safety or rights of a volunteer participating in the trial or interfere with the scientific integrity of study
* 8. Positive urine pregnancy test (HCG) on the day of vaccination

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 3 (Actual)
Dates: Start 2018-11-04 (Actual); Primary Completion 2021-10-28 (Actual); Study Completion 2021-10-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Maryland, Baltimore, Center for Vaccine Development and Global Health, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Vaccination With Oral Cholera Vaccine (Vaxchora)
Started | 3
Completed | 1
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Vaccination With Oral Cholera Vaccine (Vaxchora)
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 28 [25 to 33]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Change in the Absolute Percentage of Positive CD4+ CD25+/OX40+ T Cells
Description: Change in absolute percentage of positive CD4+ T cell (CD25+/OX40+) responses. T cell responses were defined by changes in T cell activation markers as compared to pre-immunization levels following ex vivo stimulation with cholera specific antigens. Cells were collected at baseline and on day 3 after immunization with the CVD103-HgR cholera vaccine.
Time Frame: Baseline and Day 3
Measure: Mean (Standard Deviation); unit: percentage of CD25 positive cells
Arm/Group | Vaccination With Oral Cholera Vaccine (Vaxchora)
Number analyzed (Participants) | 3
percentage of CD25 positive cells | -0.013 (0.023)

2. Primary Outcome: Change in Absolute Percentage of Positive CD4+ CD25+/OX40+ T Cells
Description: Change in absolute percentage of positive CD4+ T cell (CD25+/OX40+) responses. T cell responses were defined by changes in T cell activation markers as compared to pre-immunization levels following ex vivo stimulation with cholera specific antigens. Cells were collected at baseline and on day 5 after immunization with the CVD103-HgR cholera vaccine.
Time Frame: Baseline and Day 5
Measure: Mean (Standard Deviation); unit: percentage of CD25 positive cells
Arm/Group | Vaccination With Oral Cholera Vaccine (Vaxchora)
Number analyzed (Participants) | 3
percentage of CD25 positive cells | 0.013 (0.061)

3. Primary Outcome: Change in Absolute Percentage of Positive CD4+ CD25+/OX40+ T Cells
Description: Change in absolute percentage of positive CD4+ T cell (CD25+/OX40+) responses. T cell responses were defined by changes in T cell activation markers as compared to pre-immunization levels following ex vivo stimulation with cholera specific antigens. Cells were collected at baseline and on day 8 after immunization with the CVD103-HgR cholera vaccine.
Time Frame: Baseline and Day 8
Measure: Mean (Standard Deviation); unit: percentage of CD25 positive cells
Arm/Group | Vaccination With Oral Cholera Vaccine (Vaxchora)
Number analyzed (Participants) | 3
percentage of CD25 positive cells | 0.013 (0.050)

4. Primary Outcome: Change in Absolute Percentage of Positive CD4+ CD25+/OX40+ T Cells
Description: Change in absolute percentage of positive CD4+ T cell (CD25+/OX40+) responses. T cell responses were defined by changes in T cell activation markers as compared to pre-immunization levels following ex vivo stimulation with cholera specific antigens. Cells were collected at baseline and on day 10 after immunization with the CVD103-HgR cholera vaccine.
Time Frame: Baseline and Day 10
Measure: Mean (Standard Deviation); unit: percentage of CD25 positive cells
Arm/Group | Vaccination With Oral Cholera Vaccine (Vaxchora)
Number analyzed (Participants) | 3
percentage of CD25 positive cells | 0.153 (0.045)

5. Primary Outcome: Change in Absolute Percentage of Positive CD4+ CD25+/OX40+ T Cells
Description: Change in absolute percentage of positive CD4+ T cell (CD25+/OX40+) responses. T cell responses were defined by changes in T cell activation markers as compared to pre-immunization levels following ex vivo stimulation with cholera specific antigens. Cells were collected at baseline and on day 15 after immunization with the CVD103-HgR cholera vaccine.
Time Frame: Baseline and Day 15
Measure: Mean (Standard Deviation); unit: percentage of CD25 positive cells
Arm/Group | Vaccination With Oral Cholera Vaccine (Vaxchora)
Number analyzed (Participants) | 3
percentage of CD25 positive cells | 0.047 (0.015)

6. Primary Outcome: Change in Absolute Percentage of Positive CD4+ CD25+/OX40+ T Cells
Description: Change in absolute percentage of positive CD4+ T cell (CD25+/OX40+) responses. T cell responses were defined by changes in T cell activation markers as compared to pre-immunization levels following ex vivo stimulation with cholera specific antigens. Cells were collected at baseline and on day 29 after immunization with the CVD103-HgR cholera vaccine.
Time Frame: Baseline and Day 29
Measure: Mean (Standard Deviation); unit: percentage of CD25 positive cells
Arm/Group | Vaccination With Oral Cholera Vaccine (Vaxchora)
Number analyzed (Participants) | 3
percentage of CD25 positive cells | 0.043 (0.035)

7. Primary Outcome: Change in Absolute Percentage of Positive T Follicular/Helper 17 Cells Expressing CD154
Description: Change in absolute percentage of positive T follicular/helper 17 cells expressing CD154. T cell responses were defined by changes in T cell activation markers as compared to pre-immunization levels following ex vivo stimulation with cholera specific antigens. Cells were collected at baseline and on day 1 after immunization with the CVD103-HgR cholera vaccine.
Time Frame: Baseline and Day 1
Measure: Mean (Standard Deviation); unit: percentage of CD25 positive cells
Arm/Group | Vaccination With Oral Cholera Vaccine (Vaxchora)
Number analyzed (Participants) | 3
percentage of CD25 positive cells | 0.01 (0.01)

8. Primary Outcome: Change in Absolute Percentage of Positive T Follicular/Helper 17 Cells Expressing CD154
Description: Change in absolute percentage of positive T follicular/helper 17 cells expressing CD154. T cell responses were defined by changes in T cell activation markers as compared to pre-immunization levels following ex vivo stimulation with cholera specific antigens. Cells were collected at baseline and on day 3 after immunization with the CVD103-HgR cholera vaccine.
Time Frame: Baseline and Day 3
Measure: Mean (Standard Deviation); unit: percentage of CD25 positive cells
Arm/Group | Vaccination With Oral Cholera Vaccine (Vaxchora)
Number analyzed (Participants) | 3
percentage of CD25 positive cells | 1.06 (0.98)

9. Primary Outcome: Change in Absolute Percentage of Positive T Follicular/Helper 17 Cells Expressing CD154
Description: Change in absolute percentage of positive T follicular/helper 17 cells expressing CD154. T cell responses were defined by changes in T cell activation markers as compared to pre-immunization levels following ex vivo stimulation with cholera specific antigens. Cells were collected at baseline and on day 5 after immunization with the CVD103-HgR cholera vaccine.
Time Frame: Baseline and Day 5
Measure: Mean (Standard Deviation); unit: percentage of CD25 positive cells
Arm/Group | Vaccination With Oral Cholera Vaccine (Vaxchora)
Number analyzed (Participants) | 3
percentage of CD25 positive cells | 0.32 (0.25)

10. Primary Outcome: Change in Absolute Percentage of Positive T Follicular/Helper 17 Cells Expressing CD154
Description: Change in absolute percentage of positive T follicular/helper 17 cells expressing CD154. T cell responses were defined by changes in T cell activation markers as compared to pre-immunization levels following ex vivo stimulation with cholera specific antigens. Cells were collected at baseline and on day 8 after immunization with the CVD103-HgR cholera vaccine.
Time Frame: Baseline and Day 8
Measure: Mean (Standard Deviation); unit: percentage of CD25 positive cells
Arm/Group | Vaccination With Oral Cholera Vaccine (Vaxchora)
Number analyzed (Participants) | 3
percentage of CD25 positive cells | 0.18 (0.16)

11. Primary Outcome: Change in Absolute Percentage of Positive T Follicular/Helper 17 Cells Expressing CD154
Description: Change in absolute percentage of positive T follicular/helper 17 cells expressing CD154. T cell responses were defined by changes in T cell activation markers as compared to pre-immunization levels following ex vivo stimulation with cholera specific antigens. Cells were collected at baseline and on day 10 after immunization with the CVD103-HgR cholera vaccine.
Time Frame: Baseline and Day 10
Measure: Mean (Standard Deviation); unit: percentage of CD25 positive cells
Arm/Group | Vaccination With Oral Cholera Vaccine (Vaxchora)
Number analyzed (Participants) | 3
percentage of CD25 positive cells | 0.10 (0.18)

12. Primary Outcome: Change in Absolute Percentage of Positive T Follicular/Helper 17 Cells Expressing CD154
Description: Change in absolute percentage of positive T follicular/helper 17 cells expressing CD154. T cell responses were defined by changes in T cell activation markers as compared to pre-immunization levels following ex vivo stimulation with cholera specific antigens. Cells were collected at baseline and on day 15 after immunization with the CVD103-HgR cholera vaccine.
Time Frame: Baseline and Day 15
Measure: Mean (Standard Deviation); unit: percentage of CD25 positive cells
Arm/Group | Vaccination With Oral Cholera Vaccine (Vaxchora)
Number analyzed (Participants) | 3
percentage of CD25 positive cells | 0.27 (0.36)

13. Primary Outcome: Change in Absolute Percentage of Positive T Follicular/Helper 17 Cells Expressing CD154
Description: Change in absolute percentage of positive T follicular/helper 17 cells expressing CD154. T cell responses were defined by changes in T cell activation markers as compared to pre-immunization levels following ex vivo stimulation with cholera specific antigens. Cells were collected at baseline and on day 29 after immunization with the CVD103-HgR cholera vaccine.
Time Frame: Baseline and Day 29
Measure: Mean (Standard Deviation); unit: percentage of CD25 positive cells
Arm/Group | Vaccination With Oral Cholera Vaccine (Vaxchora)
Number analyzed (Participants) | 3
percentage of CD25 positive cells | 0.00 (0.00)

ADVERSE EVENTS:
Time Frame: approximately three years
Arm/Group | Vaccination With Oral Cholera Vaccine (Vaxchora)
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-26): https://cdn.clinicaltrials.gov/large-docs/57/NCT03724357/Prot_SAP_001.pdf